CLINICAL TRIAL: NCT00000297
Title: Effects of Labetalol on Nicotine Administration in Humans
Brief Title: Effects of Labetalol on Nicotine Administration in Humans - 14
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09259-14; P50-09259-14
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1998-10

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Labetalol

INTERVENTIONS:
Drug: Labetalol

SUMMARY:
The purpose of this study is to investigate the effects of labetalol in response to intravenous nicotine

DETAILED DESCRIPTION:
The purpose of this study is to determine whether labetalol, an alpha and beta adrenergic blocker, will block the subjective and physiological effects of intravenously administered nicotine in humans. A total of 12 subjects will participate in the double blind placebo controlled, outpatient study. Subjects will have 3 separate experimental sessions 3-9 days apart. On each of the experimental sessions, a single oral dose of low (100mg) or high dose of labetalol (200mg ), or placebo will be administered. Two hours after labetalol or placebo treatment, subjects will receive 15 variance grams nicotine base/kg intravenously. Several physiological endocrine and subjective measures will be obtained during the sessions. We propose that blockage of adrenergic receptors by labetalol will significantly block the physological and subjective effects of nicotine.

ELIGIBILITY:
Inclusion Criteria:

Male/Female, aged 21-55 years with a smoking history of at least 1 pack of cigarettes daily for at least 1 year. In good health as verified by medical history, screening examination, and screening laboratory tests.

Exclusion Criteria:

History of heart disease, peripheral vascular disease, COPD, any other medical condition which physician investigator deems inappropriate for subject participation. Pregnant or lactating or not using adequate birth control methods. Use of regular psychotropic medication (antidepressants, antipsychotics, or anxiolytics and recent psychiatric history). Chronic use of systemic steroids or antihistamines. Abuse of alcohol or any other recreational or prescription drug. Regular use of any other tobacco products, including smokeless tobacco and nicotine products.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1998-10; Study Completion 2001-12

PRIMARY OUTCOMES:
Subjective
Physiologic measures

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Gaoussou S, Attaher O, Swihart B, Traore M, Diarra S, Soumbounou IH, Ndiaye O, Issiaka D, Morrison R, Mahamar A, Duffy PE, Dicko A, Fried M. Pregnancy outcomes in a malaria-exposed Malian cohort of women of child-bearing age. Front Med (Lausanne). 2022 Dec 8;9:1061538. doi: 10.3389/fmed.2022.1061538. eCollection 2022. PMID 36569122